CLINICAL TRIAL: NCT03620201
Title: A Pilot Single Arm Open Label Trial Evaluating M7824 (Anti-PD-L1/TGF-Beta TRAP) in a Window Setting in Patients With Stage II-III HER2/Neu Positive (HER2+) Breast Cancer (BC)
Brief Title: M7824 in Treating Patients With Stage II-III HER2 Positive Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0502; NCI-2018-01184 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0502 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: interventions — bintrafusp alfa protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (M7824) (Experimental): Participants receive anti-PD-L1/TGFbetaRII fusion protein M7824 IV over 1 hour on days 1 and 15. During days 28-56 participants receive planned neoadjuvant chemotherapy.
  Interventions: Drug: Bintrafusp Alfa

INTERVENTIONS:
Drug: Bintrafusp Alfa — Given IV
  Other Names: Anti-PDL1/TGFb Trap MSB0011359C; M7824; MSB0011359C

SUMMARY:
This phase I trial studies how well anti-PD-L1/TGFbetaRII fusion protein M7824 (M7824) works in treating patients with stage II-III HER2 positive breast cancer. Immunotherapy with M7824 may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the change in tumor-infiltrating lymphocytes (TIL) percentage pre and post M7824 therapy.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of M7824 in early stage breast cancer (stage II/III).

II. To evaluate pathological response at the time of surgery after 2 doses of M7824 followed by neoadjuvant (human epidermal growth factor receptor 2) HER2 targeted therapy in combination with chemotherapy of physician's choice.

EXPLORATORY OBJECTIVES:

I. To evaluate imaging based response to M7824. II. To evaluate potential systemic and tumor based predictive biomarker candidates of response.

III. To evaluate immune responses induced by exposure to M7824 systemically and in tumor microenvironment (TME).

OUTLINE:

Patients receive anti-PD-L1/TGFbetaRII fusion protein M7824 intravenously (IV) over 1 hour on days 1 and 15. During days 28-56 patients receive planned neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and any locally-required authorization (e.g., Health Insurance Portability and Accountability Act [HIPAA]) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Tumor size >= 2 cm and with no known distant metastatic disease
* HER2+, breast cancer as defined by American Society of Clinical Oncology (ASCO)-College of American Pathologists (CAP) guidelines: HER2/neu is defined as positive: immunohistochemistry (IHC) 3+ based on circumferential membrane staining that is complete, intense in situ hybridization (ISH) positive based on: single-probe average HER2 copy number >= 6.0 signals/cell. Dual-probe HER2/CEP17 ratio >= 2.0; with an average HER2 copy number >= 4.0 signals/cell, dual-probe HER2/CEP17 ratio >= 2.0; with an average HER2, copy number < 4.0 signals/cell, dual-probe HER2/CEP17 ratio < 2.0; with an average HER2, copy number >= 6.0 signals/cell, neoadjuvant systemic therapy is planned and will include HER2 targeted therapy in combination with chemotherapy of physician's choice
* Hemoglobin >= 9 g/dL
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (>= 1500 per mm^3)
* Platelet count >= 100 x 10^9/L (>= 100,000 per mm^3)
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only upon treating physician, principal investigator (PI) or co-PI approval
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Serum creatinine clearance >= 60 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance
* Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: >= 60 years old and no menses for >= 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry and be using highly effective contraception (that is, methods with a failure rate of less than 1% per year) for both male and female subjects if the risk of conception exists (Note: The effects of the trial treatment on the developing human fetus are unknown; thus, women of childbearing potential and men must agree to use highly effective contraception). Male subjects on study must also use highly effective contraception. Highly effective contraception must be used 30 days prior to first trial treatment administration, for the duration of trial treatment, and at least for 4 months after stopping trial treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this trial, the treating physician should be informed immediately
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both EMD Serono staff and/or staff at the study site)
* Participation in another clinical study with an investigational product during the last 1 month prior to initiation of therapy
* Any previous treatment with a PD-1 or PD-L1 inhibitor or CTLA-4 inhibitor
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease >= 1 year before the first dose of study drug and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease eg, cervical cancer in situ
* Has received therapy for this current diagnosis of breast cancer including endocrine therapy or chemotherapy
* Mean QT interval corrected for heart rate (QTc) >= 470 ms
* Current or prior use of immunosuppressive medication within 28 days before the first dose of M7824, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of primary immunodeficiency
* History of organ transplants that require immunosuppression
* History of hypersensitivity to M7824 or any excipient of M7824
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses, known history of human immunodeficiency virus (HIV) and/or viral hepatitis, or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Active tuberculosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving M7824
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
* Subjects with uncontrolled seizures
* Concurrent treatment with non-permitted drugs and other interventions
* Any major surgery for any reason, except diagnostic biopsy, within 4 weeks of the enrollment
* Inflammatory breast cancer
* History of conditions associated with bleeding diatheses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Change in tumor-infiltrating lymphocytes (TIL) percentage | Baseline up to post M7824 therapy
Laboratory parameters | Up to 1 year
Eye symptoms (and signs if symptoms warranted additional evaluation) | Up to 1 year
Vital signs | Up to 1 year
Electrocardiogram parameters | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi K Murthy, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT03620201/ICF_000.pdf